CLINICAL TRIAL: NCT02247804
Title: The Efficacy and Safety of Bimatoprost SR in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Efficacy and Safety Study of Bimatoprost Sustained-Release (SR) in Participants With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 192024-091; 2014-003037-26 (EudraCT Number)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Needles; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bimatoprost SR 15 μg (Experimental): Study Eye: bimatoprost sustained release (SR) 15 μg administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Drug: Bimatoprost SR; Drug: Active Comparator: Timolol 0.5%; Other: Sham: Applicator Without Needle; Drug: Timolol Vehicle (placebo)
- Bimatoprost SR 10 μg (Experimental): Study Eye: bimatoprost SR 10 μg administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Drug: Bimatoprost SR; Drug: Active Comparator: Timolol 0.5%; Other: Sham: Applicator Without Needle; Drug: Timolol Vehicle (placebo)
- Timolol 0.5% (Active Comparator): Study Eye and Non-Study Eye: sham administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
  Interventions: Drug: Active Comparator: Timolol 0.5%; Other: Sham: Applicator Without Needle

INTERVENTIONS:
Drug: Bimatoprost SR — Bimatoprost SR administered in the study eye on Day 1, Week 16, and Week 32.
  Other Names: AGN-192024
  Arms: Bimatoprost SR 10 μg; Bimatoprost SR 15 μg
Drug: Active Comparator: Timolol 0.5% — Timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
Other: Sham: Applicator Without Needle — Sham administered on Day 1, Week 16, and Week 32.
Drug: Timolol Vehicle (placebo) — Timolol vehicle administered once in the morning and once in the evening for up to 20 months.
  Arms: Bimatoprost SR 10 μg; Bimatoprost SR 15 μg

SUMMARY:
This study will evaluate the efficacy and safety of bimatoprost SR in participants with open-angle glaucoma or ocular hypertension. The study includes a 12-month treatment period with an 8-month extended follow-up.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of either open-angle glaucoma or ocular hypertension in each eye and both eyes require IOP-lowering treatment.

Exclusion Criteria:

* Previous enrollment in another Allergan Bimatoprost SR Study.
* Eye surgery (including cataract surgery) and/or any eye laser surgery within the past 6 months in the study eye
* Anticipated need for laser eye surgery in either eye within the first 52 weeks of the study duration
* History of glaucoma surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bejanian, Study Director — Allergan
Locations (106):
- United States (56):
  - Arizona Glaucoma Specialists, Phoenix, Arizona
  - Lugene Eye Institute, Glendale, California
  - Lakeside Vision Center, Irvine, California
  - Hamilton Glaucoma Center, Shiley Eye Center UCSD, La Jolla, California
  - Atlantis Eye Care, Long Beach, California
  - Glaucoma Institute of Beverly Hills, Los Angeles, California
  - Montebello Medical Eye Center Inc., Montebello, California
  - Stanford University, Palo Alto, California
  - Foothill Eye Institute, Pasadena, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Grutzmacher, Lewis and Sierra, Inc., Sacramento, California
  - Pacific Eye Associates, San Francisco, California
  - Eye Associates of Colorado Springs, Colorado Springs, Colorado
  - Palm Beach Eye Center, INC, Atlantis, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - East Florida Eye Institute, Stuart, Florida
  - International Research Center, Tampa, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Chicago Eye Specialists, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Heart of America Eye Care PA, Shawnee Mission, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - MedRACS, LLC, Quincy, Massachusetts
  - Ocular Immunology and Uveitis Foundation, Waltham, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Eye Constultants, P.A., Bloomington, Minnesota
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Moyes Eye Center, PC, Kansas City, Missouri
  - Northern New Jersey Eye Institute P.A., South Orange, New Jersey
  - Eyecare Ophthalmology Associates, PC, Bethpage, New York
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Rochester Ophthalmological Group PC, Rochester, New York
  - 2000 North Village Avenue, Rockville Centre, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Montefiore Medical Center, The Bronx, New York
  - 8 Medical Park Drive, Asheville, North Carolina
  - Albemarle Clinical Trials, LLC, Elizabeth City, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - The Ohio State University Havener Eye Institute, Columbus, Ohio
  - Drs Fine Hoffman & Sims, LLC, Eugene, Oregon
  - Wills Eye Institute - Glaucoma Research Center, Philadelphia, Pennsylvania
  - Associates in Ophthalmology, Pittsburgh, Pennsylvania
  - Carolinas Centers for Sight PC, Florence, South Carolina
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Keystone Research, LTD, Austin, Texas
  - Glaucoma Associates of Texas, Dallas, Texas
  - The Cataract, Glaucoma & Refractive Surgery Center, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Focal Point Vision, San Antonio, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - West Virginia University, Morgantown, West Virginia
- Australia (5):
  - Vision Eye Institute Chatswood, Chatsworth
  - Melbourne Eye Specialists, Fitzroy
  - Waverley Eye Clinic, Glen Waverley
  - Marsden Eye Specialists, Parramatta, Paramatta
  - Preston Eye Clinic, Preston
- Austria (2):
  - University of Graz, Graz
  - University of Vienna, Vienna
- Belgium (2):
  - University Hospitals Leuven, Leuven
  - CHU Sart Tilman, Liège
- Brazil (7):
  - Universidade Federal de Goias, Goiânia, Goiás
  - Elo Oftalmologistas Associados, Belo Horizonte, Minas Gerais
  - Nova Campinas Oftalmologia, Campinas, São Paulo
  - Hospital Medicina dos Olhos, Osasco, São Paulo
  - Hospital de Olhos MS, Rio Verde
  - Escola Paulista de Medicina, São Paulo
  - Hospital das Clínicas - Faculdade de Medicina, São Paulo
- Glostrup Hospital, Glostrup Municipality, Denmark
- Hong Kong (2):
  - Hong Kong Eye Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong
- Hungary (3):
  - Ganglion Medical Center, Pécs
  - Markusovszky Korhaz, Szombathely
  - Zala Megyei Kórház, Zalaegerszeg
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion M.C., Haifa
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
- Centro Oftalmológico Mácula Diagnóstico y Tratamiento, Lima, Peru
- Philippines (3):
  - Asian Eye Institute, Makati
  - Pacific Eyecare & Laser Institute, Makati
  - Makati Medical Center, Makati
- Poland (9):
  - Prywatna Klinika Okulistyczna OFTALMIKA, Bydgoszcz
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Public Clinical Hospital No. 1, Lublin
  - ZOZ OKO- TEST Poradnia Okulistyczna, Nowy Targ
  - Diagnostic and Microsurgery Center of the Eye LENS, Olsztyn
  - Retina Sp. z o.o, Warsaw
  - Klinika Okulistyki WIML, Warsaw
  - Uniwersytecki Szpital Kliniczny, Warsaw
  - Uniwersyteck Szpital Kliniczny, Wroclaw
- Spain (9):
  - Institut Clinic d'Oftalmologia, Barcelona
  - Institut Catala de la Retina, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital General, Valencia
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (2):
  - Buddhist Tzu Chi General Hospital (BTCGH), Hualien City, Hualien
  - Kaohsiung Veterans General Hospital, Kaohsiung City

REFERENCES:
- [Derived] Weinreb RN, Bacharach J, Brubaker JW, Medeiros FA, Bejanian M, Bernstein P, Robinson MR. Bimatoprost Implant Biodegradation in the Phase 3, Randomized, 20-Month ARTEMIS Studies. J Ocul Pharmacol Ther. 2023 Jan-Feb;39(1):55-62. doi: 10.1089/jop.2022.0137. Epub 2022 Nov 15. PMID 36378864
- [Derived] Medeiros FA, Sheybani A, Shah MM, Rivas M, Bai Z, Werts E, Ahmed IIK, Craven ER. Single Administration of Intracameral Bimatoprost Implant 10 microg in Patients with Open-Angle Glaucoma or Ocular Hypertension. Ophthalmol Ther. 2022 Aug;11(4):1517-1537. doi: 10.1007/s40123-022-00527-6. Epub 2022 May 28. PMID 35643967
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Timolol 0.5%: Comparator: Study Eye and Non-Study Eye: sham administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
Period: Treatment Period 1
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started | 198 | 198 | 198
Received (Sham or Bimatoprost SR) | 193 | 197 | 197
Completed | 176 | 194 | 190
Not Completed | 22 | 4 | 8
Not completed — Adverse Event | 9 | 2 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Personal Reasons | 7 | 1 | 2
Not completed — Protocol Deviation | 0 | 0 | 1
Not completed — Randomized but not Treated | 5 | 1 | 1
Period: Treatment Period 2
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 172 | 191 | 187
Completed | 164 | 186 | 179
Not Completed | 8 | 5 | 8
Not completed — Adverse Event | 6 | 3 | 3
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Personal Reasons | 2 | 1 | 1
Not completed — Reason not Specified | 0 | 0 | 2
Period: Treatment Period 3
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Started (Started=received administration (Sham or Bimatoprost SR) in the cycle) | 158 | 183 | 177
Completed | 147 | 173 | 167
Not Completed | 11 | 10 | 10
Not completed — Adverse Event | 4 | 3 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Personal Reasons | 4 | 3 | 2
Not completed — Reason not Specified | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population was defined as all randomized participants.
Groups:
- Bimatoprost SR 15 μg: Study Eye: bimatoprost SR 15 μg administered on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol vehicle administered once in the morning and once in the evening for up to 20 months. Non-Study Eye: sham administration on Day 1 (Period 1), Week 16 (Period 2), and Week 32 (Period 3); timolol 0.5% administered once in the morning and once in the evening for up to 20 months.
- Total: Total of all reporting groups
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator | Total
Number analyzed (Participants) | 198 | 198 | 198 | 594
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (13.0) | 62.6 (11.5) | 62.5 (11.0) | 62.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 86 | 106 | 288
  Male | 102 | 112 | 92 | 306
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 122 | 123 | 130 | 375
  Black or African American | 30 | 31 | 21 | 82
  Asian | 12 | 17 | 16 | 45
  Hispanic | 27 | 23 | 25 | 75
  Other | 6 | 4 | 5 | 15
  Not Reported | 1 | 0 | 1 | 2
Intraocular Pressure (IOP) [Mean (Full Range); unit: mm Hg] — IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye.
  mm Hg
    Hour 0 | 24.76 [18.0 to 32.0] | 24.64 [21.5 to 32.0] | 24.63 [16.0 to 32.0] | 24.68 [16.0 to 32.0]
    Hour 2 | 23.56 [19.0 to 32.0] | 23.29 [19.0 to 32.0] | 23.19 [16.0 to 32.0] | 23.35 [16.0 to 32.0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in IOP in the Study Eye at Week 12 (Hours 0 and 2)
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. A mixed-effects model with repeated measures (MMRM) was used for analyses. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline (Hours 0 and 2) to Week 12 (Hours 0 and 2)
Population: ITT population was defined as all randomized participants. Number analyzed is the number of participants with evaluable data at the given timepoint.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mm Hg)
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 198 | 198 | 198
millimeters of mercury (mm Hg)
  Change from Baseline at Hour 0, Week 12: number analyzed (Participants) | 185 | 192 | 191
  Change from Baseline at Hour 0, Week 12 | -6.46 (0.29) | -6.38 (0.28) | -6.05 (0.28)
  Change from Baseline at Hour 2, Week 12: number analyzed (Participants) | 183 | 192 | 191
  Change from Baseline at Hour 2, Week 12 | -7.18 (0.26) | -6.69 (0.25) | -6.48 (0.25)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 12, Hour 0: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — MMRM analyses was used with response variable:IOP time-matched change from baseline;Fixed factors: Treatment,timepoint,treatment-by-timepoint interaction and baseline IOP stratification;Covariate:Time-matched baseline IOP and timepoint by time-matched baseline IOP interaction. Unstructured covariance matrix was used; p = 0.2950, MMRM; Least-squares Mean Difference = -0.41, 95% CI 2-sided [-1.17 to 0.36], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 12, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3904, MMRM; Least-squares Mean Difference = -0.33, 95% CI 2-sided [-1.09 to 0.43], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 12, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0464, MMRM; Least-squares Mean Difference = -0.70, 95% CI 2-sided [-1.40 to -0.01], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 12, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Week 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5383, MMRM; Least-squares Mean Difference = -0.21, 95% CI 2-sided [-0.90 to 0.47], Standard Error of Mean 0.35

2. Primary Outcome: IOP in the Study Eye at Week 2 (Hour 0)
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. MMRM was used for analyses.
Time Frame: Week 2 (Hour 0)
Population: ITT population was defined as all randomized participants. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 191 | 196 | 196
mm Hg | 16.82 (0.25) | 17.02 (0.25) | 17.83 (0.25)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 2, Hour 0: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0033, MMRM; Least-squares Mean Difference = -1.01, 95% CI 2-sided [-1.68 to -0.34], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 2, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0187, MMRM; Least-squares Mean Difference = -0.80, 95% CI 2-sided [-1.47 to -0.13], Standard Error of Mean 0.34

3. Primary Outcome: IOP in the Study Eye at Week 2 (Hour 2)
Description: as for outcome 2
Time Frame: Week 2 (Hour 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 191 | 196 | 196
mm Hg | 16.48 (0.22) | 16.42 (0.22) | 17.33 (0.22)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 2, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0057, MMRM; Least-squares Mean Difference = -0.85, 95% CI [-1.45 to -0.25], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 2, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0031, MMRM; Least-squares Mean Difference = -0.90, 95% CI [-1.50 to -0.31], Standard Error of Mean 0.30

4. Primary Outcome: IOP in the Study Eye at Week 6 (Hour 0)
Description: as for outcome 2
Time Frame: Week 6 (Hour 0)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 188 | 197 | 194
mm Hg | 17.08 (0.24) | 16.88 (0.23) | 17.71 (0.24)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 6, Hour 0: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0547, MMRM; Least-squares Mean Difference = -0.63, 95% CI [-1.26 to 0.01], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 6, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0107, MMRM; Least-squares Mean Difference = -0.82, 95% CI [-1.46 to -0.19], Standard Error of Mean 0.32

5. Primary Outcome: IOP in the Study Eye at Week 6 (Hour 2)
Description: as for outcome 2
Time Frame: Week 6 (Hour 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 187 | 197 | 193
mm Hg | 16.62 (0.23) | 16.51 (0.22) | 17.16 (0.23)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 6, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0860, MMRM; Least-squares Mean Difference = 0.08, 95% CI [-1.16 to 0.08], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 6, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0362, MMRM; Least-squares Mean Difference = -0.66, 95% CI [-1.27 to -0.04], Standard Error of Mean 0.31

6. Primary Outcome: IOP in the Study Eye at Week 12 (Hour 0)
Description: as for outcome 2
Time Frame: Week 12 (Hour 0)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 185 | 192 | 191
mm Hg | 17.53 (0.29) | 17.61 (0.28) | 17.94 (0.28)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 12, Hour 0: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2950, MMRM; Least-squares Mean Difference = -0.41, 95% CI [-1.17 to 0.36], Standard Error of Mean 0.39
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 12, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3904, MMRM; Least-squares Mean Difference = -0.33, 95% CI 2-sided [-1.09 to 0.43], Standard Error of Mean 0.39

7. Primary Outcome: IOP in the Study Eye at Week 12 (Hour 2)
Description: as for outcome 2
Time Frame: Week 12 (Hour 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 183 | 192 | 191
mm Hg | 16.81 (0.26) | 17.30 (0.25) | 17.51 (0.25)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Week 12, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0464, MMRM; Least-squares Mean Difference = -0.70, 95% CI [-1.40 to -0.01], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Week 12, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared non-inferior to timolol 0.5% if the upper limit of the 95% CI was ≤ 1.5 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5383, MMRM; Least-squares Mean Difference = -0.21, 95% CI [-0.90 to 0.47], Standard Error of Mean 0.35

8. Secondary Outcome: Change From Baseline in IOP in the Study Eye
Description: IOP is a measurement of the fluid pressure inside the study eye. Measurements were taken at Hours 0 and 2. The study eye is defined as the eye that meets the entry criteria. If both eyes meet the entry criteria, the eye with the higher IOP at Baseline Hour 0 will be selected as the study eye. If both eyes had the same IOP at Hour 0, then the right eye was designated as the study eye. MMRM was used for analyses. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time Frame: Baseline (Hours 0 and 2) to Weeks 2 and 6 (Hours 0 and 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
Number analyzed (Participants) | 198 | 198 | 198
mm Hg
  Change from Baseline at Hour 0, Week 2: number analyzed (Participants) | 191 | 196 | 196
  Change from Baseline at Hour 0, Week 2 | -7.17 (0.25) | -6.97 (0.25) | -6.17 (0.25)
  Change from Baseline at Hour 2, Week 2: number analyzed (Participants) | 191 | 196 | 196
  Change from Baseline at Hour 2, Week 2 | -7.52 (0.22) | -7.57 (0.22) | -6.67 (0.22)
  Change from Baseline at Hour 0, Week 6: number analyzed (Participants) | 188 | 197 | 194
  Change from Baseline at Hour 0, Week 6 | -6.91 (0.24) | -7.11 (0.23) | -6.29 (0.24)
  Change from Baseline at Hour 2, Week 6: number analyzed (Participants) | 187 | 197 | 193
  Change from Baseline at Hour 2, Week 6 | -7.37 (0.23) | -7.48 (0.22) | -6.83 (0.23)
Statistical Analysis 1: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 2, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0033, MMRM; Least-squares Mean Difference = -1.01, 95% CI 2-sided [-1.68 to -0.34], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0187, MMRM; Least-squares Mean Difference = -0.80, 95% CI 2-sided [-1.47 to -0.13], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 2, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0057, MMRM; Least-squares Mean Difference = -0.85, 95% CI 2-sided [-1.45 to -0.25], Standard Error of Mean 0.31
Statistical Analysis 4: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 2, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0031, MMRM; Least-squares Mean Difference = -0.90, 95% CI 2-sided [-1.50 to -0.31], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 6, Hour 0: The null hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0547, MMRM; Least-squares Mean Difference = -0.63, 95% CI 2-sided [-1.26 to 0.01], Standard Error of Mean 0.32
Statistical Analysis 6: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 6, Hour 0: The null hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0107, MMRM; Least-squares Mean Difference = -0.82, 95% CI 2-sided [-1.46 to -0.19], Standard Error of Mean 0.32
Statistical Analysis 7: Comparison: Bimatoprost SR 15 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 6, Hour 2: The null hypothesis was that bimatoprost SR 15 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0860, MMRM; Least-squares Mean Difference = -0.54, 95% CI 2-sided [-1.16 to 0.08], Standard Error of Mean 0.32
Statistical Analysis 8: Comparison: Bimatoprost SR 10 μg vs Timolol 0.5%: Comparator; Change from Baseline Week 6, Hour 2: The null hypothesis was that bimatoprost SR 10 μg was to be declared superior to timolol 0.5% if the upper limit of the 95% CI was < 0 mm Hg for all scheduled timepoints (Hours 0 and 2 at Weeks 2, 6, 12); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0362, MMRM; Least-squares Mean Difference = -0.66, 95% CI [-1.27 to -0.04], Standard Error of Mean 0.31

ADVERSE EVENTS:
Time Frame: First dose of study drug to last visit (Up to approximately 20 months)
Description: Safety population included all participants who received at least 1 dose of study treatment.
Arm/Group | Bimatoprost SR 15 μg | Bimatoprost SR 10 μg | Timolol 0.5%: Comparator
All-Cause Mortality (participants affected / at risk) | 2/193 | 1/197 | 1/197
Serious Adverse Events (participants affected / at risk) | 31/193 | 25/197 | 18/197
Other Adverse Events (participants affected / at risk) | 143/193 | 138/197 | 105/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost SR 15 μg (N=193) | Bimatoprost SR 10 μg (N=197) | Timolol 0.5%: Comparator (N=197)
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Corneal endothelial cell loss (Eye disorders) | 12 | 4 | 0
Corneal oedema (Eye disorders) | 3 | 2 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0
Corneal touch (Eye disorders) | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 1 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Internal haemorrhage (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost SR 15 μg (N=193) | Bimatoprost SR 10 μg (N=197) | Timolol 0.5%: Comparator (N=197)
Conjunctival hyperaemia (Eye disorders) | 74 | 60 | 47
Foreign body sensation in eyes (Eye disorders) | 31 | 23 | 12
Eye pain (Eye disorders) | 28 | 26 | 12
Eye irritation (Eye disorders) | 28 | 18 | 22
Photophobia (Eye disorders) | 23 | 19 | 4
Corneal endothelial cell loss (Eye disorders) | 20 | 14 | 0
Conjunctival haemorrhage (Eye disorders) | 19 | 17 | 16
Iritis (Eye disorders) | 19 | 11 | 1
Dry eye (Eye disorders) | 17 | 19 | 12
Punctate keratitis (Eye disorders) | 16 | 12 | 14
Lacrimation increased (Eye disorders) | 13 | 10 | 12
Vision blurred (Eye disorders) | 12 | 10 | 11
Corneal oedema (Eye disorders) | 12 | 5 | 2
Anterior chamber cell (Eye disorders) | 11 | 9 | 0
Nasopharyngitis (Infections and infestations) | 13 | 10 | 14
Influenza (Infections and infestations) | 8 | 13 | 4
Intraocular pressure increased (Investigations) | 13 | 20 | 7
Headache (Nervous system disorders) | 8 | 14 | 7
Visual field defect (Nervous system disorders) | 4 | 10 | 5
Hypertension (Vascular disorders) | 17 | 12 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT02247804/SAP_000.pdf
  • Study Protocol (2017-03-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT02247804/Prot_001.pdf